CLINICAL TRIAL: NCT07218042
Title: Are Two Needles Really Better Than One? A Time, Economic, and Environmental Evaluation of EBUS-TBNA
Brief Title: Study of Procedural Efficiency in EBUS With Dual Versus Single NEEDLEs: Evaluating the Value of a Second Needle in EBUS as it Pertains to Economic and Environmental Impact
Acronym: SPEED NEEDLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Kapp (Other)
Collaborators: Duke University (Other); University of California, Davis (Other)
Responsible Party: Sponsor-Investigator, Christopher Kapp, Assistant Professor of Medicine, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STU00220729
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Mediastinal and Hilar Lymphadenopathy
Keywords: Bronchoscopy; EBUS

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- One EBUS Needle (Active Comparator): Patients underwent a standard of care EBUS with one needle utilized in the procedure.
  Interventions: Diagnostic Test: We randomized patients to the two arms above; there was no specific intervention performed other than randomizing patients to one or two needles.
- Two EBUS Needle (Experimental): Patients underwent standard of care EBUS with two needles used.
  Interventions: Diagnostic Test: We randomized patients to the two arms above; there was no specific intervention performed other than randomizing patients to one or two needles.

INTERVENTIONS:
Diagnostic Test: We randomized patients to the two arms above; there was no specific intervention performed other than randomizing patients to one or two needles. — We randomized patients to the two arms above; there was no specific intervention performed other than randomizing patients to one or two needles.

SUMMARY:
Currently, the EBUS bronchoscopy procedure uses either one or two needles to perform the biopsy of the lymph node based on physician preference. We want to determine the optimal number of needles to use for future EBUS bronchoscopy procedures like the one you are scheduled to have for your care and investigate the economic and environmental impact and time involved in using one versus two needles.

DETAILED DESCRIPTION:
Endobronchial Ultrasound (EBUS) is a mainstay of diagnostic bronchoscopy, as it is performed for mediastinal and hilar lymph node sampling for cancer staging, diagnosis of sarcoidosis, lymphoma, infection, and other disease processes. It is a procedure that is commonplace in all bronchoscopy suites across the world.

In our bronchoscopy suite, our current practice varies based on the bronchoscopist and number of lymph nodes requiring sampling in a procedure (can range from 1-5) as to whether one or two needles are utilized. The bronchoscopist may use two needles to save time when multiple lymph nodes must be biopsied or if an individual node needs to be biopsied several times to obtain more tissue for pathologic study.

EBUS needles are single use and there is one randomized trial (n=20 patients) that showed a decreased time of procedure in patients where two needles were used versus one (Khan et al., 2013). However, no data exist evaluating the economic impact (cost of needle versus endoscopy dollars saved) or environmental impact of using one versus two needles. This study will examine these factors to determine the optimal way to perform this procedure in the future, considering the procedure and anesthesia time, economic costs, and environmental costs.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a bronchoscopy with lymph node sampling

Exclusion Criteria:

* Unable to get a bronchoscopy procedure for various reasons
* Other criteria per protocol uploaded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time Under Anesthesia | During bronchoscopy procedure

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT07218042/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT07218042/ICF_001.pdf